CLINICAL TRIAL: NCT02707887
Title: Technology Enhanced Behavioral Activation Treatment for Substance Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-0815; R01DA026424 (NIH)
Record Dates: First submitted 2015-05-27; First posted 2016-03-14 (Estimated); Last update posted 2023-10-16 (Actual); Status verified 2021-01

CONDITIONS: Substance-Related Disorders; Depressive Disorder; Behavioral Symptoms; Risk-Taking; Sexual Behavior
Keywords: Mental Disorders; Mood Disorders; Behavioral Activation
MeSH Terms: conditions — Substance-Related Disorders; Depressive Disorder; Behavioral Symptoms; Risk-Taking; Sexual Behavior; Mental Disorders; Mood Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment as Usual (Placebo Comparator): Patients are offered substance use group therapy including relapse prevention. They are also provided medical consultation on an ongoing basis as needed.
  Interventions: Behavioral: Treatment as Usual
- LETS ACT (Active Comparator): The Life Enhancement Treatment for Substance Use (LETS ACT) involves the discussion of the treatment rationale, identification of values and goals in various life areas and activities in line with chosen life areas, and training for patients to identify their cycle of negative mood and behavior using forms to track their daily goals.
  Interventions: Behavioral: LETS ACT; Behavioral: Treatment as Usual
- LETS ACT-SE (Active Comparator): Participants assigned to the smartphone-enhanced LETS ACT (LETS ACT-SE) condition will be provided the exact same treatment as outlined in LETS ACT, except that LETS ACT-SE participants will record their daily goals using smartphone technology.
  Interventions: Behavioral: LETS ACT-SE; Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: LETS ACT — The Life Enhancement Treatment for Substance Use (LETS ACT)
  Other Names: Behavioral Activation; Life Enhancement Treatment for Substance Use
  Arms: LETS ACT
Behavioral: LETS ACT-SE — Participants assigned to the smartphone-enhanced LETS ACT (LETS ACT-SE) condition will be provided the exact same treatment as outlined in LETS ACT, except that LETS ACT-SE participants will record their daily goals using smartphone technology.
  Other Names: Behavioral Activation; Smartphone-Enhanced LETS ACT
  Arms: LETS ACT-SE
Behavioral: Treatment as Usual — Participants will receive the treatment typically provided to patients at the substance use treatment facility.
  Other Names: TAU

SUMMARY:
The purpose of this study is to:

1. test the effect of a smartphone enhanced LETS ACT (LETS ACT-SE) on frequency of substance use
2. use functional magnetic resonance imaging (fMRI) to test the relationship between neuromarkers of reward sensitivity on frequency of substance use.

DETAILED DESCRIPTION:
Comorbid substance use disorder (SUD) and depression is highly prevalent and associated with elevated rates of post treatment relapse to substance use, HIV risk behavior, and associated poor mental and physical health outcomes. Further, rates of substance use and depression disproportionately affect minority groups and those living in poverty. Although efficacious, the often complex, specialized nature of CBT poses problems in its integration into substance use treatment programs. Budget cuts for mental health and substance use treatment both nationally and in the state of North Carolina, reduce availability of publically funded treatment programs and staff to patient ratios. To address this limitation, a behavioral activation (BA) treatment, the Life Enhancement Treatment for Substance Use (LETS ACT), was developed to treat depressive symptoms among a predominantly African American sample of low income illicit drug users currently receiving residential substance use treatment. Collectively, two Stage I studies and 1 year follow-up data from the investigators Stage II R01DA026424 indicate that compared to a control condition, LETS ACT is associated with significantly better outcomes for treatment retention, post treatment abstinence, HIV sexual risk behavior, depressive symptoms, and environmental reward.

Although these strong outcomes suggest that LETS ACT may be ready for a Stage III dissemination trial, it is of note that there was a significant indirect effect of LETS ACT homework compliance on post treatment substance use and HIV sexual risk behavior via the theoretically proposed BA mechanism of action, environmental reward. In the context of limited access to care, these findings point to the need to identify cost-effective delivery-vehicles to increase treatment engagement outside of clinician sessions. Further, identifying neuroscience based biomarkers (neuromarkers) underlying key theoretical aspects of BA (i.e., reward sensitivity), and their relation to heterogeneity in BA treatment response among substance users with depression, are critical for the identification of accurately targeted interventions.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 55
* Meet criteria for DSM-V substance use disorder
* Elevated depressive symptoms (BDI ≥ 14)

Exclusion Criteria:

* Limited mental competency (MMSE < 23)
* Psychosis
* The use of psychotropic medication for < 3 months
* The inability to give informed, voluntary, written consent to participate

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 206 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Timeline Followback (TLFB) | TLFB will be assessed from baseline to a 12-month follow up period.
  The Time Line Follow Back is a self-report measure of drug and alcohol use.

SECONDARY OUTCOMES:
Behavioral Activation for Depression Scale (BADS) | BADS will be assessed from baseline to a 12-month follow up period.
  The BADS is a 25-item self-report measure of overall level of activity involvement
Reward Probability Index (RPI) | RPI will be assessed from baseline to a 12-month follow up period.
  The RPI is a 20-item self-report measure used to assess environmental reward and punishment.
Beck Depression Inventory-II (BDI-II) | BDI-II will be evaluated from baseline to a 12-month follow up period
  The Beck Depression Inventory is a 21-item self-report measure of depressive symptoms
Daily Goals Form | Baseline to a 3-months post treatment.
  The Daily Goals Form is used to measure Treatment Engagement.
Texas Christian University (TCU) HIV/AIDS Risk Assessment Form | TCU will be assessed from baseline to a 12-month follow up period.
  The TCU is a self-structured interview that measures HIV risk behavior in the domains of drug use and sex
Urinalysis | Urinalysis is assessed from post treatment to a 12-month follow up period
  Urinalysis is a biological measure of substance use.
Breathalyzer | Breathalyzer will be assessed from baseline to a 12-month follow up period.
  Breathalyzer is a biological measure of alcohol use.
Short Form Health Survey (SF-12) | SF-12 will be assessed from baseline to a 12-month follow up period.
  The SF-12 is a 12-item self-report measure of mental and physical health-related functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Daughters, Ph.D., Principal Investigator — University of North Carolina
Locations (2):
- United States (2):
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Southlight Healthcare, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kane L, Reese ED, Paquette C, Paladino M, Linares Abrego P, Daughters SB. Substance use negatively impacts change in reinforcement during the year following substance use treatment. Psychol Addict Behav. 2025 May;39(3):238-253. doi: 10.1037/adb0001051. Epub 2025 Jan 9. PMID 39786834
- [Derived] Paquette CE, Rubalcava DT, Chen Y, Anand D, Daughters SB. A Mobile App to Enhance Behavioral Activation Treatment for Substance Use Disorder: App Design, Use, and Integration Into Treatment in the Context of a Randomized Controlled Trial. JMIR Form Res. 2021 Nov 3;5(11):e25749. doi: 10.2196/25749. PMID 34730535